CLINICAL TRIAL: NCT01824251
Title: NPB-01(Intravenous Immunoglobulin) Maintenance Therapy for Patients With Chronic Inflammatory Demyelinating Polyneuropathy.
Brief Title: Phase III Clinical Trial of NPB-01maintenance Therapy in Patients With Chronic Inflammatory Demyelinating Polyneuropathy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPB-01-09/C-01
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: IVIG in Chronic Inflammatory Demyelinating Polyneuropathy; Patients with Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPB-01 (Experimental): Intravenous immunoglobulin
  Interventions: Drug: NPB-01

INTERVENTIONS:
Drug: NPB-01
  Other Names: Intravenous immunoglobulin

SUMMARY:
Patients diagnosed with Chronic Inflammatory Demyelinating Polyneuropathy were confirmed based on the European Federation of Neurological Societies/ Peripheral. Nerve Society Guideline. Patients who meet all inclusion criteria and do not conflict with the exclusion criteria will receive NPB-01 (intravenous immunoglobulin) 400mg/kg/day for five consecutive days. Subsequently, patients receive NPB-01 1g/kg every 3weeks and evaluate the Inflammatory Neuropathy Cause and Treatment（INCAT） score and INCAT sensory sumscore（ISS） et al.

As a safety endpoint, the safety of NPB-01 will be investigated the occurrence of adverse events by one year after the start of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with progressive or relapsing motor and sensory dysfunction of more than one limb resulting from neuropathy within 2 months prior to the date informed consent is obtained.
* 2. Patients who INCAT score between 2-9. (If the INCAT score is 1 in upper limb, the INCAT score of 2 must be exclusively from leg disability to qualify.)
* 3. Patients who need high-dose intravenous immunoglobulin therapy.
* 4. Patients who continued treatment for CIDP without addition or increase at 30 days before informed consent.
* 5. Patients with greater than or equal to twenty years old at informed consent.

Exclusion Criteria:

* 1. Patients with evidence of myelopathy or demyelination of central nerve
* 2. Patients with evidence of stroke, central nerve system trauma, or persistent neurological deficits due to peripheral neuropathy from other causes（diabetic neuropathy, IgM paraproteinaemia, uraemic neuropathy, toxic neuropathy, hereditary neuropathy）
* 3. Patients with evidence of neuropathy or alcoholic neuropathy or vitamin deficiency neuropathy due to myeloma, lymphoma, sarcoidosis, systemic lupus erythematosus, malignancy, vasculitis, Crow-Fukase syndrome, Sjögren syndrome.
* 4. Patients with multifocal motor neuropathy.
* 5. Patients treated with plasmapheresis at 3 months before informed consent.
* 6. Patients treated with rituximab at 6 months before informed consent.
* 7. Patients treated with high-dose intravenous immunoglobulin（greater than or equal to 1g/kg） at 8 weeks before informed consent.
* 8. Patients treated with intravenous immunoglobulin at 3 weeks before informed consent.
* 9. Patients with history of shock or hypersensitivity for NPB-01.
* 10. Patients with IgA deficiency.
* 11. Patients with malignancy at informed consent.
* 12. Patients with impaired liver function.
* 13. Patients with impaired renal function.
* 14. Patients with cerebro- or cardiovascular disorders.
* 15. Patients with high risk of thromboembolism.
* 16. Patients with hemolytic/hemorrhagic anemia.
* 17. Patients with decreased cardiac function.
* 18. Patients with decreased platelet.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
proportion of patients with more than 1point improvement in the INCAT score relative to baseline at 28weeks. | 28weeks
proportion of patients with more than 1point exacerbation in the INCAT score relative to 28weeks at 52weeks. | 52weeks

SECONDARY OUTCOMES:
INCAT score | 1,4,7,10,13,16,19,22,25,28,31,34,37,40,43,46,49,52weeks
ISS | 1,4,7,10,13,16,19,22,25,28,31,34,37,40,43,46,49,52weeks
maximum grip strength | 1,4,7,10,13,16,19,22,25,28,31,34,37,40,43,46,49,52weeks
Medical Research Council（MRC） sum score | 1,4,7,10,13,16,19,22,25,28,31,34,37,40,43,46,49,52weeks
the amplitude of the compound muscle action potential of the most severely affected motor nerve | 1,4,28,52weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon Pharmaceutical Co., Ltd, Osaka, Japan

REFERENCES:
- [Derived] Kuwabara S, Mori M, Misawa S, Suzuki M, Nishiyama K, Mutoh T, Doi S, Kokubun N, Kamijo M, Yoshikawa H, Abe K, Nishida Y, Okada K, Sekiguchi K, Sakamoto K, Kusunoki S, Sobue G, Kaji R; Glovenin-I CIDP Study Group. Intravenous immunoglobulin for maintenance treatment of chronic inflammatory demyelinating polyneuropathy: a multicentre, open-label, 52-week phase III trial. J Neurol Neurosurg Psychiatry. 2017 Oct;88(10):832-838. doi: 10.1136/jnnp-2017-316427. Epub 2017 Aug 2. PMID 28768822